CLINICAL TRIAL: NCT03450759
Title: An Open-label, Randomized, Four-way Cross-over, Single Oral Dose Study Comparing the Pharmacokinetics of Four Different Formulations of AZD9977 (Part A) and Influence of Food (Part B) in Healthy Male Subjects
Brief Title: A Single Oral Dose Study to Evaluate Four Different Formulations of AZD9977 and the Effect of Food in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D6401C00002
Record Dates: First submitted 2018-02-15; First posted 2018-03-01 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Healthy Volunteers
Keywords: Heart failure.; Mineralocorticoid receptor modulator.; Heart failure with preserved ejection fraction (HFpEF).
MeSH Terms: conditions — Heart Failure | interventions — AZD9977

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment sequence 1 (Experimental): In Part A, randomized subjects will receive orally single dose of all treatments in fasted condition in the following sequence:
  AZD9977 oral suspension (reference) AZD9977 capsule AZD9977 ER capsule (fast rate) AZD9977 ER capsule (Int. rate)
  Interventions: Drug: AZD9977 Oral suspension (reference); Drug: AZD9977 capsule; Drug: AZD9977 ER capsule (fastvrate); Drug: AZD9977 ER capsule (Int. rate)
- Treatment sequence 2 (Experimental): In Part A, randomized subjects will receive orally single dose of all treatments in fasted condition in the following sequence:
  AZD9977 capsule AZD9977 ER capsule (fast rate) AZD9977 ER capsule (Int. rate) AZD9977 oral suspension (reference)
  Interventions: Drug: AZD9977 Oral suspension (reference); Drug: AZD9977 capsule; Drug: AZD9977 ER capsule (fastvrate); Drug: AZD9977 ER capsule (Int. rate)
- Treatment sequence 3 (Experimental): In Part A, randomized subjects will receive orally single dose of all treatments in fasted condition in the following sequence:
  AZD9977 ER capsule (fast rate) AZD9977 ER capsule (Int. rate) AZD9977 Oral suspension (reference) AZD9977 capsule
  Interventions: Drug: AZD9977 Oral suspension (reference); Drug: AZD9977 capsule; Drug: AZD9977 ER capsule (fastvrate); Drug: AZD9977 ER capsule (Int. rate)
- Treatment sequence 4 (Experimental): In Part A, randomized subjects will receive orally single dose of all treatments in fasted condition in the following sequence:
  AZD9977 ER capsule (Int. rate) AZD9977 Oral suspension (reference) AZD9977 capsule AZD9977 ER capsule (fast rate)
  Interventions: Drug: AZD9977 Oral suspension (reference); Drug: AZD9977 capsule; Drug: AZD9977 ER capsule (fastvrate); Drug: AZD9977 ER capsule (Int. rate)

INTERVENTIONS:
Drug: AZD9977 Oral suspension (reference) — Randomized subjects will receive single oral dose of AZD9977 oral suspension 15 mg/mL on Days 1, 3, 5 and 7 in Part A.
Drug: AZD9977 capsule — Randomized subjects will receive single oral dose of AZD9977 capsule 65 mg on Days 1, 3, 5 and 7 in Part A.
Drug: AZD9977 ER capsule (fastvrate) — Randomized subjects will receive single oral dose of AZD9977 ER capsule (fast rate) 65 mg on Days 1, 3, 5 and 7 in Part A.
Drug: AZD9977 ER capsule (Int. rate) — Randomized subjects will receive single oral dose of AZD9977 ER capsule (Int rate) 65 mg on Days 1, 3, 5 and 7 in Part A.

SUMMARY:
This study will evaluate pharmacokinetics (PK) of four different formulations with different release profiles of AZD9977 (PART A) in the fasted state, and one of the formulation will be selected for further development (Part B). In Part B, the influence of food on the PK of AZD9977 will be evaluated

DETAILED DESCRIPTION:
This study is a randomized, open-label, single-center study conducted on 12 healthy male subjects. This consists of three periods:

* Screening period (only prior to Day-1)
* Residential/treatment period (Part A and Part B)
* Follow-up period (5 to 7 days after-final dose)

The study is divided into 2 parts: Part A and B. The subjects will participate in both Part A and Part B. Part A will be a 4-way cross-over study to compare the PK of 3 different solid formulations with different release rates with an oral suspension of AZD9977 in fasting conditions. Subjects in Part A will receive the following treatments on Days 1, 3, 5 and 7:

* AZD9977 oral suspension 15 mg/mL (15 mg/mL = 195 mg) (reference)
* AZD9977 capsule, 65 mg (3 x 65 mg = 195 mg)
* AZD9977 extended release (ER) capsule, 65 mg, fast (3 x 65 mg = 195 mg)
* AZD9977 ER capsule, 65 mg, intermediate release (Int) (3 x 65 mg = 195 mg) Subjects will be resident from 1 day before Part A until at least 36 hours post last dosing in Part A. Subjects will return to the unit for Part B after completion of Part A. There will be a washout period of at least 2 days between the doses for a subject. Based on the results in Part A, one of the solid formulations will be selected and evaluated in fed conditions on Day of Part B. Subjects will return to the unit for a final study visit 5 to 7 days post- dose in Part B. Each subject will be involved in the study for approximately 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male subjects aged 18 to 50 years with suitable veins for cannulation or repeated venipuncture.
3. Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
4. Provision of signed, written and dated informed consent for optional genetic research. If a subject decline to participate in the genetic component of the study, there will be no penalty or loss of benefit to the subject. The subject will not be excluded from other aspects of the study described in this protocol.
5. Subject judged likely to complete and agree to eat a specified high-fat, high-calorie standardized FDA breakfast.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the PI, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
2. History or presence of gastrointestinal (GI), hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
4. Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, as judged by the PI including: Serum potassium > 5.0 mmol/L
5. Any clinically significant abnormal findings in vital signs as specified below and as judged by the PI at screening and on admission: Systolic blood pressure (SBP) < 90 mmHg or > 140 mmHg; Diastolic blood pressure (DBP) < 50 mmHg or > 90 mmHg; Heart rate (HR) < 45 or > 90 beats per minute (bpm)
6. Any clinically significant abnormalities on 12-lead ECG, as judged by the PI.
7. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.
8. Known or suspected history of drug abuse in the last 12 months, as judged by the PI.
9. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose or 1 month after the last visit whichever is the longest. Note: subjects consented and screened, but not randomized in this study or a previous Phase 1 study, are not excluded.
10. Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
11. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to AZD9977.
12. Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 3 months prior to screening.
13. Positive screen for drugs of abuse, cotinine or alcohol at screening or on each admission to the study center.
14. Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
15. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life.
16. Known or suspected history of alcohol or drug abuse or excessive intake of alcohol in the last 12 months as judged by the PI.
17. Involvement of any AstraZeneca, PAREXEL or study site employee or their close relatives
18. Subjects who have previously received AZD9977.
19. Judgment by the PI that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
20. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
21. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection or previous bone marrow transplant.
22. Subjects with any special dietary restrictions such as subjects that are lactose intolerant or are vegetarians/vegans.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability (Frel) of AZD9977 capsule, ER (fast rate) and ER (Int. rate) capsules versus AZD9977 oral suspension (reference): Area under plasma concentration-time curve from time zero to infinity (AUC) | Dosing sessions: Part A: Days 1, 3, 5 and 7; Part B: Day 1
  To assess Frel by assessments of PK parameters AUC after administration of single oral dose of AZD9977 capsule and ER (fast rate and Int. rate) capsules by comparison with AZD9977 oral suspension (reference).
Relative bioavailability (Frel) of AZD9977 capsule, ER (fast rate) and ER (Int. rate) capsules versus AZD9977 oral suspension (reference): Area under the plasma concentration-curve from time zero to time of last quantifiable concentration (AUClast) | Dosing sessions: Part A: Days 1, 3, 5 and 7; Part B: Day 1
  To assess Frel by assessments of PK parameters AUClast after administration of single oral dose of AZD9977 capsule and ER (fast rate and Int. rate) capsules by comparison with AZD9977 oral suspension (reference).
Relative bioavailability (Frel) of AZD9977 capsule, ER (fast rate) and ER (Int. rate) capsules versus AZD9977 oral suspension (reference): Area under the plasma concentration-time curve from time zero to time 24 hours (AUC[0-24]) | Dosing sessions: Part A: Days 1, 3, 5 and 7; Part B: Day 1
  To assess Frel by assessments of PK parameters AUC[0-24] after administration of single oral dose of AZD9977 capsule and ER (fast rate and Int. rate) capsules by comparison with AZD9977 oral suspension (reference).
Relative bioavailability (Frel) of AZD9977 capsule, ER (fast rate) and ER (Int. rate) capsules versus AZD9977 oral suspension (reference): Maximum observed plasma concentration (Cmax ) | Dosing sessions: Part A: Days 1, 3, 5 and 7; Part B: Day 1
  To assess Frel by assessments of PK parameters Cmax after administration of single oral dose of AZD9977 capsule and ER (fast rate and Int. rate) capsules by comparison with AZD9977 oral suspension (reference).
Plasma PK parameter: Area under plasma concentration-time curve from time zero to infinity (AUC) | Dosing sessions: Part A: Days 1, 3, 5 and 7; Part B: Day 1
  To assess AUC after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Plasma PK parameter: Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUClast) | Dosing sessions: Part A: Days 1, 3, 5 and 7; Part B: Day 1
  To assess AUClast after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Plasma PK parameter: Maximum observed plasma concentration (Cmax) | Dosing sessions: Part A: Days 1, 3, 5 and 7; Part B: Day 1
  To assess Cmax after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Plasma PK parameter: Area under the plasma concentration-time curve from time zero to time 24 hours (AUC[0-24]) | Dosing sessions: Part A: Days 1, 3, 5 and 7
  To assess AUC(0-24) after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
The Effect of food on the PK of one of the solid formultaion evaluated in Part A under fasting and fed conditions in Part B | Dosing sessions: Part A: Days 1, 3, 5 and 7; Part B: Day 1
  To evaluate the influence of food by comparing AUC and Cmax under fasting and fed conditions for one of the solid formulations evaluated in Part A.

SECONDARY OUTCOMES:
Plasma PK parameter: Plasma concentration 24 hours post-dose (C4) | Dosing sessions: Part A and Part B - Day 1 (24 hours post-dose)
  To assess C24 after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Plasma PK parameter: Time to reach maximum observed plasma concentration (tmax) | Dosing sessions: Part A: Days 1, 3, 5 and 7; Part B: Day 1
  To assess tmax after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Plasma PK parameter: Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t½λz ) | Dosing sessions: Part A: Days 1, 3, 5 and 7; Part B: Day 1
  To assess t½λz after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Plasma PK parameter: Mean residence time of the unchanged drug in the systemic circulation from zero to infinity (MRT) | Dosing sessions: Part A: Days 1, 3, 5 and 7; Part B: Day 1
  To assess MRT after administration of single oral dose of AZD9977 capsule, ER (fast rate and Int. rate) capsules and oral suspension (reference).
Plasma PK parameter: Terminal elimination rate constant (λz) | Dosing sessions: Part A: Days 1, 3, 5 and 7; Part B: Day 1
  To assess λz after administration of single oral dose of AZD9977 capsule, ER (fast rate and Int. rate) capsules and oral suspension (reference).
Plasma PK parameter: Apparent total body clearance of drug from plasma after extravascular administration AZD9977 (CL/F) | Dosing sessions: Part A: Days 1, 3, 5 and 7; Part B: Day 1
  To assess CL/F after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Plasma PK parameter: Apparent volume of distribution during the terminal phase after extravascular administration AZD9977 (Vz/F) | Dosing sessions: Part A: Days 1, 3, 5 and 7; Part B: Day 1
  To assess Vz/F after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Number of subjects with adverse events (AEs) due to AZD9977 | From screening up to follow-up (5 to 7 days after final dose)
  To assess AEs as variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference). AEs will be collected from the start of screening throughout the treatment period up to and including the follow-up visit. Serious AEs will be recorded from the time of informed consent.
Vital sign: Blood pressure [BP] | From screening up to follow-up (5 to 7 days after final dose)
  To assess supine position systolic and diastolic BP as variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference). Both SBP and DBP will be collected after the subject has rested in the supine position for at least 5 minutes.
Vital sign: Pulse rate | From screening up to follow-up (5 to 7 days after final dose)
  To assess supine position pulse rate as variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference). Pulse rate will be collected after the subject has rested in the supine position for at least 5 minutes.
Number of participants with abnormal findings in Resting 12-lead Electrocardiogram (ECG) | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess any clinically significant abnormalities in the cardiovascular system functioning using a 10-second 12-lead ECG as variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference). The specific type and nature of the abnormality will be documented in ClinBase. Clinically significant findings will also be documented on the AE page of the CRF if applicable.
Number of participants with abnormal physical examination findings | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess any clinically significant abnormal physical examination findings as a variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference). Brief physical examination includes assessment of the general appearance, skin, abdomen, cardiovascular system and respiratory. Full physical examination includes assessment of the general appearance, respiratory, cardiovascular, abdomen, skin, head, and neck (including ears, eyes, nose, and throat), lymph nodes, thyroid, musculoskeletal and neurological systems.
Laboratory assessments: Hematology - Blood cells count | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess red blood cells ( RBC) and white blood cells (WBC) countas a variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Laboratory assessments: Hematology - Hemoglobin (Hb) | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess Hb as a variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Laboratory assessments: Hematology - Hematocrit (HCT) and Reticulocyte absolute count | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess HCT (RBC) and reticulocyte absolute count (immature RBCs) as a variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Laboratory assessments: Hematology - Mean corpuscular volume (MCV) | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess MCV as a variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Laboratory assessments: Hematology - Mean corpuscular hemoglobin (MCH) | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess MCH as a variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Laboratory assessments: Hematology - Mean corpuscular hemoglobin concentration (MCHC) | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess MCHC as a variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Laboratory assessments: Hematology - Differential count | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess differential WBC count (absolute count of neutrophils, lymphocytes, monocyets, eosinophils and basophils) as a variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Laboratory assessments: Hematology - Platelets | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess platelets count as a variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Laboratory assessments: Serum Clinical chemistry - sodium, potassium, calcium and phosphate | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess serum sodium, potassium, calcium and phosphate level as a variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Laboratory assessments: Serum Clinical chemistry - Urea and Uric acid | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess serum urea and uric acid level as a variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Laboratory assessments: Serum Clinical chemistry - Creatinine | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess serum creatinine level as a variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Laboratory assessments: Serum Clinical chemistry - Albumin | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess serum albumin level as a variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Laboratory assessments: Serum Clinical chemistry - Glucose (fasting) | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess serum fasting glucose level as a variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Laboratory assessments: Serum Clinical chemistry - C-reactive protein (CRP) | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess serum CRP level as a variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Laboratory assessments: Serum Clinical chemistry - Liver enzymes | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess serum Alkaline phosphatase (ALP), Alanine aminotransferase (ALT), Aspartate aminotransferase (AST) and Gamma glutamyl transpeptidase (GGT) level as a variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Laboratory assessments: Serum Clinical chemistry - Bilirubin | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess serum bilirubin (total and unconjugated) level as a variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Laboratory assessments: Serum Clinical chemistry - High-sensitivity troponin T | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess serum high-sensitivity troponin T level as a variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Laboratory assessments: Serum Clinical chemistry - Creatine kinase | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess serum creatine kinase level as a variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Laboratory assessments: Serum Clinical chemistry - N-terminal-pro-brain natriuretic peptide (NT-proBNP) | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess serum NT-proBNP level as a variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Laboratory assessments: Clinical Urinalysis - Glucose | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess urine glucose level as a variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference).
Laboratory assessments: Clinical Urinalysis - Protein | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess urine protein level as a variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference). If urinalysis is positive for protein, a microscopy test will be performed to assess RBC, WBC, casts [cellular, granular, hyaline]).
Laboratory assessments: Clinical Urinalysis - Blood | At screening, dosing sessions of Part A and Part B and follow-up (5 to 7 days after final dose)
  To assess presence of blood in urine as a variable of safety and tolerability after administration of single oral dose of AZD9977 capsule, ER capsules (fast rate and Int. rate) and oral suspension (reference). If urinalysis is positive for blood, a microscopy test will be performed to assess RBC, WBC, casts [cellular, granular, hyaline]).

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No